CLINICAL TRIAL: NCT02479321
Title: Efficacy of Goal Directed Hemodynamic Therapy Based on Noninvasive Monitoring to Reduce Perioperative Complications in Patients With Hip Fracture
Brief Title: Goal Directed Hemodynamic Therapy Based on Noninvasive Monitoring in Patients With Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juan-Víctor Lorente, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Juan-Víctor Lorente, MD, PhD, Medical Doctor, Althaia Xarxa Assistencial Universitària de Manresa
Organization: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIC 15/03
Record Dates: First submitted 2015-06-15; First posted 2015-06-24 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Hip Fractures
Keywords: Fluid therapy; Aged; Perioperative complications; Survival; Intraoperative Goal Directed Therapy
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Hemodynamic optimization according to the standards of perioperative monitoring of our center. In the intraoperative period hemodynamic monitoring will be done by management of blood pressure, heart rate and oxygen saturation
- GDT noninvasive monitoring group (Experimental): GDT based on noninvasive monitoring System ClearSight® and Platform EV Clinic 1000®
  Interventions: Other: GDT based on noninvasive monitoring; Device: System ClearSight® and Platform EV Clinic 1000®

INTERVENTIONS:
Other: GDT based on noninvasive monitoring — Before entering the operating room, hemodynamic optimization start by optimizing preload with Fluid Challenge according to evidence-based GDT protocols. Once stabilized the cardiovascular system after induction of anesthesia, hemodynamic optimization continue with Mini Fluid Challenge.
  In the intraoperative period, hemodynamic optimization is based on maintaining systolic blood pressure and stroke volume. A Mini Fluid Challenge is administered to patients who respond to volume or a vasoactive drug according cardiac index for non-responders.
  Other Names: Intraoperative Goal-Directed Hemodynamic Therapy
  Arms: GDT noninvasive monitoring group
Device: System ClearSight® and Platform EV Clinic 1000® — Hemodynamic control is held by non-invasive continuous monitoring techniques (system ClearSight® and Platform EV Clinic 1000®). Monitored variables: blood pressure, heart rate, oxygen saturation, cardiac output, cardiac index, stroke volume and stroke volume index.
  Arms: GDT noninvasive monitoring group

SUMMARY:
Crude incidence rate in Spain of hip fracture in people over 65 years was 511 cases per 100,000 in 2002. About 30% of patients die in the first year. Cardiocirculatory complications during and after surgery partly explain this high morbidity and mortality. Most patients are frail and with multicomorbidity. Goal-Directed Hemodynamic Therapy (GDT) based on noninvasive continuous monitoring of blood pressure, heart rate, oxygen saturation, cardiac output, cardiac index, stroke volume and stroke volume index can reduce perioperative complications and improve survival. The objective of our study is to assess the efficacy of a goal-directed hemodynamic therapy in reducing perioperative complications. Patients and Methods: non-randomized intervention study with a historical control and 1-year follow-up. Patients older than 64 years with non-traumatic hip fracture requiring surgical intervention. In the control group standard care was performed based on non-invasive, intermittent arterial pressure measurement, obtained every 5 minutes, continuous heart rate, and oxygen saturation. In the intervention group GDT based on noninvasive monitoring will be performed. The main outcome will be the percentage of patients with perioperative complications. Secondary outcomes: LOS and survival at 12 months of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture that require surgical treatment
* Agree to participate and sign informed consent

Exclusion Criteria:

* Pathological or traffic related fractures
* Anesthetic contraindication for surgery
* Refractures
* Contraindication for hemodynamic monitoring
* Physiocal less than 30 after 7 minutes
* Psychomotor agitation that prevents hemodynamic monitoring

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 568 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who developed intraoperative haemodynamic instability | Intraoperative period
  Intraoperative haemodynamic instability, defined as one measurement of SAP < 90 mmHg in the CG and for at least one minute in the IG and/or the need for a bolus of vasoconstrictor.

SECONDARY OUTCOMES:
Intraoperative arrhythmias | Intraoperative period
  Electrocardiographic evidence of cardiac rhythm disturbance.
Postoperative complications | Postoperative period
  Major cardiovascular complications, minor cardiovascular complications, Respiratory, Renal, Infections, Surgical reintervention during hospital stay
Hospital stay | Patients will be followed for the duration of hospital stay, an expected median of 11 days
  Length of hospital stay (days)
Survival | One-year survival

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bosch Sabater, MD PhD, Study Chair — Althaia Xarxa Assistencial Universitària de Manresa; Francesca Reguant Corominas, MD PhD, Study Chair — Althaia Xarxa Assistencial Universitària de Manresa
Locations (1):
- Althaia Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona, Spain

REFERENCES:
- [Derived] Lorente JV, Reguant F, Arnau A, Borderas M, Prieto JC, Torrallardona J, Carrasco L, Solano P, Perez I, Farre C, Jimenez I, Ripolles-Melchor J, Monge MI, Bosch J. Effect of goal-directed haemodynamic therapy guided by non-invasive monitoring on perioperative complications in elderly hip fracture patients within an enhanced recovery pathway. Perioper Med (Lond). 2022 Aug 10;11(1):46. doi: 10.1186/s13741-022-00277-w. PMID 35945605